CLINICAL TRIAL: NCT05700240
Title: Effect of Orthokeratology on Myopia Progression in French Children
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Professeur Jean-Baptiste CONART, Professeur, Central Hospital, Nancy, France
Other Study IDs: 2022PI090
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Myopia Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Orthokeratology treatment
  Interventions: Device: orthokeratology
- single-vision spectacle correction
  Interventions: Device: single-vision spectacle correction

INTERVENTIONS:
Device: orthokeratology — rigid contact lenses
  Groups: Orthokeratology treatment
Device: single-vision spectacle correction — simple wear of spectacle
  Groups: single-vision spectacle correction

SUMMARY:
To evaluate and to compare the effect of orthokeratology (OK) on axial elongation in French myopic children.

ELIGIBILITY:
Inclusion Criteria:

* 7 to 17 years old
* Myopia between 0,50 D and 7.00 D
* Astigmatism ≤ 4.00 D with-the-rule 180+-20
* Anisometropia ≤ 1.50 D
* Myopia evolution ≥ 0.25 D over 6 months
* Best-corrected visual acuity (BCVA) ≥ 20/20 (Snellen equivalent)
* Follow-up period > 6 months

Exclusion Criteria:

* Prior history of any other myopia control treatment (except for single vision distance spectacles)
* Contraindication for contact lens wear or orthokeratology
* Preexisting ocular (amblyopia, strabismus, ocular inflammation, trauma, or surgery) or systemic disease
* Poor compliance to lens wear, examination or follow-up

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 64 consecutive myopic children who underwent OK treatment or single-vision spectacle correction at a private ophthalmology clinic in Nancy from November 2019 to December 2020
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-11-02 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Changes in axial length at one year | one year

SECONDARY OUTCOMES:
changes in refractive error | one year
changes in choroidal thickness | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Jean-Baptiste CONART, Nancy, France